CLINICAL TRIAL: NCT02399020
Title: Social Cognition and Interaction Training (SCIT) for Adults With Psychotic Disorder: An Open Pilot Study in Finland
Brief Title: Social Cognition and Interaction Training for Adults With Psychotic Disorders: An Open Pilot Study in Finland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); City of Helsinki (Other)
Responsible Party: Principal Investigator, Jorma Oksanen MD, chief physician, Jorvi Psychosis Clinic, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 169/13/03/03/2011
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Psychotic Disorder; Cognitive Function 1, Social
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCIT group (Experimental): Social Cognition and Interaction Training intervention group
  Interventions: Behavioral: Social Cognition and Interaction Training

INTERVENTIONS:
Behavioral: Social Cognition and Interaction Training — manualized group treatment providing training in facial emotion recognition, understanding the role of emotion in social situations, training with videoed vignettes to avoid jumping to conclusions in order to avoid attributional biases, tolerating ambiguity and distinguishing facts from guesses, skill consolidation and generalization to everyday life situations.

SUMMARY:
33 individuals with a psychotic disorder were given 22-24 sessions weekly or twice weekly of Social Cognition and Interaction Training (SCIT) and evaluated at the baseline and after the intervention. Main outcome was improvement in social cognition according to specific measures of facial emotion identification, Theory of Mind, attributional bias, social cognitive accuracy and metacognitive overconfidence.

DETAILED DESCRIPTION:
33 clinically stable in- and outpatients with chart diagnoses of schizophrenia, schizoaffective disorder or unspecified nonorganic psychosis, aged 18-56 years, were given 22-24 weekly or twice weekly sessions of a manualized group treatment for improvement of social cognition, Social Cognition and Interaction Training (1,2). Main outcome was defined as improvement in social cognition according to specific measures of facial emotion identification, Theory of Mind, attributional bias, social cognitive accuracy and metacognitive overconfidence.Emotion perception was measured with the Facial Emotion Identification Task (FEIT) (3); Theory of Mind was measured with the Hinting Task (4) and attributional bias with the Ambiguous Intentions Hostility Questionnaire-Ambiguous Items (AIHQ-A) (5). In addition, broad-based social cognitive accuracy, attributional bias and metacognitive overconfidence was measured with the Social Cognition Screening Questionnaire. All the measures were evaluated at the baseline and immediately after the intervention. Changes in total scores for the FEIT and Hinting Task, and the three subscales of AIHQ-A and SCSQ were analysed separately using paired samples t-test in IBM SPSS Statistics version 21.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of schizophrenia, schizoaffective disorder or psychosis NOS
* inpatients in longer-stay rehabilitation wards or outpatients in supported housing
* stable clinical condition
* written informed consent
* problems in social relationships according to the clinical staff
* standard medical treatment provided by the care facilities

Exclusion Criteria:

* inadequate command of Finnish language
* unstable clinical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
improvement in social cognitive ability | 11-24 weeks
  improvement according to measures of facial emotion recognition, theory of mind, attributional bias and social cognitive accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Leena Turpeinen, MD, Study Director — City of Helsinki Department of Social Services and Health Care
Locations (1):
- Aurora Hospital, Helsinki, Finland

REFERENCES:
- [Background] Roberts DL, Penn DL. Social cognition and interaction training (SCIT) for outpatients with schizophrenia: a preliminary study. Psychiatry Res. 2009 Apr 30;166(2-3):141-7. doi: 10.1016/j.psychres.2008.02.007. Epub 2009 Mar 9. PMID 19272654
- [Background] Penn DL, Roberts DL, Combs D, Sterne A. Best practices: The development of the Social Cognition and Interaction Training program for schizophrenia spectrum disorders. Psychiatr Serv. 2007 Apr;58(4):449-51. doi: 10.1176/ps.2007.58.4.449. PMID 17412842
- [Background] Kerr SL, Neale JM. Emotion perception in schizophrenia: specific deficit or further evidence of generalized poor performance? J Abnorm Psychol. 1993 May;102(2):312-8. doi: 10.1037//0021-843x.102.2.312. PMID 8315144
- [Background] Corcoran R, Mercer G, Frith CD. Schizophrenia, symptomatology and social inference: investigating "theory of mind" in people with schizophrenia. Schizophr Res. 1995 Sep;17(1):5-13. doi: 10.1016/0920-9964(95)00024-g. PMID 8541250
- [Background] Combs DR, Penn DL, Wicher M, Waldheter E. The Ambiguous Intentions Hostility Questionnaire (AIHQ): a new measure for evaluating hostile social-cognitive biases in paranoia. Cogn Neuropsychiatry. 2007 Mar;12(2):128-43. doi: 10.1080/13546800600787854. PMID 17453895